CLINICAL TRIAL: NCT03907319
Title: Retrospective Multi-Site Re-Evaluation of the MRI Defined STN and Its Correlation to Motor Outcomes With Stimulation Treatment
Brief Title: SIS Evaluation of the MRI Defined Subthalamic Nucleus*
Acronym: STN
Status: Terminated | Type: Observational
Why Stopped: Enrollment not sufficient for data analysis.
Sponsor: Surgical Information Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SIS DOC-0013
Record Dates: First submitted 2019-04-02; First posted 2019-04-08 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Deep Brain Stimulation
Keywords: STN; Parkinson's Disease; Subthalamic Nucleus
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: SIS System — Software technology for visualization of anatomical structures in the brain

SUMMARY:
Retrospective review of images used to target the STN during DBS procedure and ability of the Surgical Information Sciences ("SIS") system to visualize the STN location.

DETAILED DESCRIPTION:
The purpose of this study is to collect retrospective data to demonstrate the ability of the SIS system to visualize the MRI-defined STN in patients with Parkinson's Disease (PD) who have undergone deep brain stimulation (DBS) procedure targeting the STN.

ELIGIBILITY:
Key Inclusion Criteria:

* Idiopathic PD
* Bilateral or unilateral STN-HFS for PD
* 40% improvement response to medications preoperatively

Key Exclusion Criteria:

* Missing required MR/CT imaging data

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have completed bilateral or unilateral high frequency stimulation of the subthalamic nucleus (STN-HFS) for idiopathic PD and have pre and post operative MR and CT imaging, programming data, Unified Parkinson's Disease Rating Scale Part III (UPDRS-III) scores and a 3-6 month follow-up evaluation
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Percent of STN Visualization Success | Day 1
  Measure the proportion of images successfully processed for visualization of the STN over total number of image sets
Incidence of DBS Lead Location in Proximity to STN | Day 1
  Determine incidence in which the location of the DBS lead is in or outside the STN

SECONDARY OUTCOMES:
Rate of Correlation of Predicted Outcome to Monopolar Review Outcome | 1 Month
  Rate of blinded predicted outcome compared to monopolar review outcomes
Rate of Correlation of DBS Lead Location to Long Term Outcomes | 3-6 months
  Rate of agreement between SIS-defined model of STN and actual DBS lead location and clinical motor outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Noam Harel, PhD, Principal Investigator — Surgical Information Sciences
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No